CLINICAL TRIAL: NCT02477332
Title: A Multi-center, Randomized, Double-blind, Placebo, and Active-controlled Phase 2b Dose-finding Study of QGE031 as add-on Therapy to Investigate the Efficacy and Safety in Patients With Chronic Spontaneous Urticaria (CSU)
Brief Title: Dose-finding Study of QGE031 as add-on Therapy to Evaluate Efficacy and Safety in Patients With CSU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQGE031C2201; 2014-005559-16 (EudraCT Number)
Record Dates: First submitted 2015-06-11; First posted 2015-06-22 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2018-10

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: QGE031; ligelizumab; omalizumab; chronic; spontaneous; urticaria; adults; CSU
MeSH Terms: conditions — Chronic Urticaria; Bronchiolitis Obliterans Syndrome; Urticaria | interventions — ligelizumab; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- QGE031 24 mg s.c. q4w (Experimental): ligelizumab 24 mg injection subcutaneous every 4 weeks
  Interventions: Biological: QGE031
- QGE031 72 mg s.c. q4w (Experimental): ligelizumab 72 mg injection subcutaneous every 4 weeks
  Interventions: Biological: QGE031
- QGE031 240 mg s.c. q4w (Experimental): ligelizumab 240 mg injection subcutaneous every 4 weeks
  Interventions: Biological: QGE031
- Omalizumab 300 mg s.c. q4w (Active Comparator): omalizumab 300 mg injection subcutaneous every 4 weeks
  Interventions: Biological: Omalizumab
- Placebo s.c. q4w (Placebo Comparator): placebo injection subcutaneous every 4 weeks
  Interventions: Other: Placebo
- QGE031 120 mg s.c. s.d. (Experimental): ligelizumab 120 mg injection subcutaneous single dose
  Interventions: Biological: QGE031

INTERVENTIONS:
Biological: QGE031
  Arms: QGE031 120 mg s.c. s.d.; QGE031 24 mg s.c. q4w; QGE031 240 mg s.c. q4w; QGE031 72 mg s.c. q4w
Biological: Omalizumab
  Arms: Omalizumab 300 mg s.c. q4w
Other: Placebo
  Arms: Placebo s.c. q4w

SUMMARY:
This is a placebo and active-controlled phase 2b dose-finding study to evaluate efficacy and safety of QGE031 monthly subcutaneous injections as add-on therapy in patients with Chronic Spontaneous Urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic spontaneous urticaria for at least 6 months
* Diagnosis of chronic spontaneous urticaria refractory to standard of care at time of randomization

Exclusion Criteria:

* Clearly defined underlying etiology for chronic urticaria other than chronic spontaneous urticaria
* Evidence of parasitic infection
* Any other skin disease with chronic itching
* Previous treatment with omalizumab or QGE031
* Contraindications to or hypersensitivity to fexofenadine, loratadine, cetirizine, or epinephrine
* History of anaphylaxis
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for patients participating in the study
* History of hypersensitivity to any of the study drugs or its components of similar chemical classes
* Pregnant or nursing (lactating) women

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2017-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (77):
- United States (25):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Forest Hills, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Lake Oswego, Oregon
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Katy, Texas
  - Novartis Investigative Site, South Burlington, Vermont
  - Novartis Investigative Site, Spokane, Washington
- Australia (5):
  - Novartis Investigative Site, Campbelltown, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, East Melbourne, Victoria
- Canada (3):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Québec
- Germany (7):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
- Greece (3):
  - Novartis Investigative Site, Haidari Athens, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
- Japan (11):
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
- Russia (5):
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
- Spain (12):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Taiwan (3):
  - Novartis Investigative Site, Taoyuan District, Taiwan
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- United Kingdom (3):
  - Novartis Investigative Site, Yeovil, Somerset
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Metz M, Bernstein JA, Gimenez-Arnau AM, Hide M, Maurer M, Sitz K, Soong W, Sussman G, Hua E, Barve A, Barbier N, Balp MM, Severin T. Ligelizumab improves angioedema, disease severity and quality-of-life in patients with chronic spontaneous urticaria. World Allergy Organ J. 2022 Nov 15;15(11):100716. doi: 10.1016/j.waojou.2022.100716. eCollection 2022 Nov. PMID 36440464
- [Derived] Maurer M, Gimenez-Arnau A, Bernstein JA, Chu CY, Danilycheva I, Hide M, Makris M, Metz M, Savic S, Sitz K, Soong W, Staubach P, Sussman G, Barve A, Burciu A, Hua E, Janocha R, Severin T. Sustained safety and efficacy of ligelizumab in patients with chronic spontaneous urticaria: A one-year extension study. Allergy. 2022 Jul;77(7):2175-2184. doi: 10.1111/all.15175. Epub 2021 Nov 22. PMID 34773261
- [Derived] Maurer M, Gimenez-Arnau AM, Sussman G, Metz M, Baker DR, Bauer A, Bernstein JA, Brehler R, Chu CY, Chung WH, Danilycheva I, Grattan C, Hebert J, Katelaris C, Makris M, Meshkova R, Savic S, Sinclair R, Sitz K, Staubach P, Wedi B, Loffler J, Barve A, Kobayashi K, Hua E, Severin T, Janocha R. Ligelizumab for Chronic Spontaneous Urticaria. N Engl J Med. 2019 Oct 3;381(14):1321-1332. doi: 10.1056/NEJMoa1900408. PMID 31577874
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 574 subjects screened; 382 subjects randomized; 338 (88.5%) subjects completed treatment epoch; 349 (91.4%) subjects entered follow-up phase and 320 (83.8%) completed the follow-up epoch
Period: Overall Study
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo s.c. q4w | QGE031 120 mg s.c. s.d.
Started | 43 | 84 | 85 | 85 | 43 | 42
Completed | 40 | 77 | 73 | 72 | 39 | 37
Not Completed | 3 | 7 | 12 | 13 | 4 | 5
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 1 | 2
Not completed — Lack of Efficacy | 1 | 2 | 1 | 2 | 1 | 1
Not completed — Non-compliance with study treatment | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 3 | 3 | 1 | 1
Not completed — Technical problems | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized patients, removing misrandomized patients provided that study drug was not administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo s.c. q4w | QGE031 120 mg s.c. s.d. | Total
Number analyzed (Participants) | 43 | 84 | 85 | 85 | 43 | 42 | 382
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 77 | 85 | 81 | 41 | 37 | 360
  >=65 years | 4 | 7 | 0 | 4 | 2 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (14.36) | 44.3 (12.38) | 42.9 (10.51) | 41.8 (13.06) | 45.4 (11.22) | 42.4 (14.54) | 43.3 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 61 | 67 | 66 | 31 | 30 | 286
  Male | 12 | 23 | 18 | 19 | 12 | 12 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Hives Response (HSS7=0)
Description: The primary objective was to establish the dose-response relationship of ligelizumab (24, 72 and 240 mg every 4 weeks) with respect to achievement of complete hives response (HSS7=0) at Week 12 and select an appropriate dose (or range of doses) which is likely to be superior to omalizumab at the highest approved dose (300 mg every 4 weeks).
  Hives Severity Score (HSS) is on a scale of 0 to 3. A weekly score (HSS7) is derived by adding up the average daily scores of the preceding 7 days, with a possible range of 0 - 21.
  Hives Severity Score scale:
  0 - None
  1. - Mild (1-6 hives/12 hours)
  2. - Moderate (7-12 hives/12 hours)
  3. - Severe (>12 hives/12 hours)
  To confirm an overall dose-response signal based on MCP-Mod, and to estimate the minimal ligelizumab dose that shows a relevant superior effect over omalizumab, based on the selected dose response model, the lowest ligelizumab dose that provides a response rate 15% higher than the response of omalizumab 300 mg.
Time Frame: Week 12
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo s.c. q4w | QGE031 120 mg s.c. s.d.
Number analyzed (Participants) | 43 | 84 | 85 | 85 | 43 | 42
Percentage of participants | 30.2 [17.2 to 46.1] | 51.2 [40.0 to 62.3] | 42.4 [31.7 to 53.6] | 25.9 [17.0 to 36.5] | 0 [0.0 to 8.2] | 19.0 [8.6 to 34.1]
Statistical Analysis 1: Comparison: QGE031 24 mg s.c. q4w vs QGE031 72 mg s.c. q4w vs QGE031 240 mg s.c. q4w vs Omalizumab 300 mg s.c. q4w; Test type: Superiority; p < .05, Regression, Logistic; Target dose was based on this estimated dose response. The 60% CI included the 20 - 80th percentile of target dose estimated in the bootstrap samples; Estimated target dose = 32.5, 60% CI 2-sided [27.5 to 42.5] — Min dose with effect size >15%

2. Secondary Outcome: Complete Hives Response (HSS7=0) Rate at Week 12 Measured Over 7 Days
Description: Hives Severity Score (HSS) is on a scale of 0 to 3. A weekly score (HSS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 to 21.
  Complete hives response defined as HSS7 = 0.
  Hives Severity Score scale:
  0 - None
  1. - Mild (1-6 hives/12 hours)
  2. - Moderate (7-12 hives/12 hours)
  3. - Severe (>12 hives/12 hours)
Time Frame: Week 12
Population: Full analysis set (FAS) included all randomized patients, removing misrandomized patients provided that study drug was not administered. As per protocol and SAP, for the efficacy endpoints at Week 12 or Week 20, only the QGE031 24, 72 & 240 mg, omalizumab 300 mg and placebo arms were analyzed for efficacy comparison between treatment groups.
Measure: Number; unit: Particpants
Groups:
- Placebo: placebo injection subcutaneous every 4 week
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 43 | 84 | 85 | 85 | 43
Particpants | 13 | 43 | 36 | 22 | 0

3. Secondary Outcome: Change From Baseline in Hives Severity Score (HSS7) at Week 12 Measured Over 7 Days
Description: Hives Severity Score (HSS) is on a scale of 0 to 3. A weekly score (HSS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 to 21.
  Hives Severity Score scale:
  0 - None
  1. - Mild (1-6 hives/12 hours)
  2. - Moderate (7-12 hives/12 hours)
  3. - Severe (>12 hives/12 hours)
Time Frame: Week 12
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 40 | 81 | 78 | 77 | 41
Score on a scale | -9.75 [-15.75 to -2.50] | -15.50 [-20.00 to -6.00] | -13.50 [-19.00 to -9.00] | -11.00 [-16.50 to -4.50] | -6.50 [-13.00 to -2.33]

4. Secondary Outcome: HSS7=0 Response: at Week 20 Measured Over 7 Days
Description: as for outcome 2
Time Frame: Week 20
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 43 | 84 | 85 | 85 | 43
Participants | 11 | 43 | 38 | 29 | 4

5. Secondary Outcome: Change From Baseline in Hives Severity Score (HSS7) at Week 20 Measured Over 7 Days
Description: as for outcome 3
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 39 | 78 | 74 | 73 | 40
Score on a scale | -9.00 [-12.50 to -3.50] | -16.50 [-20.50 to -6.83] | -14.00 [-19.50 to -9.00] | -11.00 [-16.00 to -4.25] | -7.50 [-13.50 to -2.25]

6. Secondary Outcome: Change From Baseline in Itch Severity Score (ISS7) at Week 12 Measured Over 7 Days
Description: Itch Severity Score (ISS) is on a scale of 0 to 3. A weekly score (ISS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 to 21.
  Itch Severity Score scale:
  0 - None
  1. - Mild (minimal awareness, easily tolerated)
  2. - Moderate (definite awareness, bothersome but tolerable)
  3. - Severe (difficult to tolerate)
Time Frame: Week 12
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 40 | 81 | 78 | 77 | 41
Score on a scale | -7.50 [-12.75 to -3.50] | -9.50 [-14.50 to -6.00] | -9.00 [-14.00 to -4.50] | -8.00 [-11.50 to -4.50] | -5.50 [-8.50 to -2.50]

7. Secondary Outcome: Change From Baseline in Itch Severity Score (ISS7) at Week 20 Measured Over 7 Days
Description: as for outcome 6
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 39 | 78 | 74 | 73 | 40
Score on a scale | -7.00 [-11.00 to -2.00] | -10.25 [-14.00 to -6.50] | -10.00 [-14.00 to -5.50] | -8.83 [-11.50 to -3.50] | -5.00 [-9.50 to -2.25]

8. Secondary Outcome: Change From Baseline in Urticaria Activity Score (UAS7) at Week 12 Measured Over 7 Days
Description: UAS7 is the sum of the HSS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42.
Time Frame: Week 12
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 40 | 81 | 78 | 77 | 41
Score on a scale | -19.50 [-26.75 to -6.25] | -26.50 [-33.00 to -12.00] | -21.75 [-32.50 to -14.00] | -19.00 [-29.00 to -8.50] | -12.00 [-21.00 to -6.00]

9. Secondary Outcome: Change From Baseline in Urticaria Activity Score (UAS7) at Week 20 Measured Over 7 Days
Description: UAS7 is the sum of the HSS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42.
Time Frame: Week 20
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Score on a scale
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 39 | 78 | 74 | 73 | 40
Score on a scale | -16.00 [-23.00 to -7.00] | -27.00 [-33.00 to -15.00] | -22.92 [-32.50 to -13.50] | -18.50 [-28.50 to -11.00] | -13.00 [-21.00 to -5.50]

10. Secondary Outcome: Complete Urticaria Activity Score Response (UAS7=0) Rate at Week 12 Measured Over 7 Days
Description: UAS7 is the sum of the HSS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42.
  Complete urticaria activity response is defined as UAS7 = 0.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 43 | 84 | 85 | 85 | 43
Participants | 13 | 37 | 34 | 22 | 0

11. Secondary Outcome: UAS7=0 Response: at Week 20 Measured Over 7 Days
Description: as for outcome 10
Time Frame: Week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 43 | 84 | 85 | 85 | 43
participants | 8 | 33 | 34 | 26 | 2

12. Secondary Outcome: Complete Itch Response (ISS7=0) Rate at Week 12 Measured Over 7 Days
Description: Itch Severity Score (ISS) is on a scale of 0 to 3. A weekly score (ISS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 to 21.
  Complete itch response defined as ISS7 = 0.
  Itch Severity Score scale:
  0 - None
  1. - Mild (minimal awareness, easily tolerated)
  2. - Moderate (definite awareness, bothersome but tolerable)
  3. - Severe (difficult to tolerate)
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 43 | 84 | 85 | 85 | 43
participants | 17 | 40 | 36 | 25 | 2

13. Secondary Outcome: ISS7=0 Response: at Week 20 Measured Over 7 Days
Description: as for outcome 12
Time Frame: Week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo
Number analyzed (Participants) | 43 | 84 | 85 | 85 | 43
participants | 8 | 35 | 36 | 28 | 3

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 44 weeks.
Arm/Group | QGE031 24 mg s.c. q4w | QGE031 72 mg s.c. q4w | QGE031 240 mg s.c. q4w | Omalizumab 300 mg s.c. q4w | Placebo s.c. q4w | QGE031 120 mg s.c. s.d.
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/84 | 0/85 | 0/85 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 3/43 | 2/84 | 2/85 | 3/85 | 4/43 | 4/42
Other Adverse Events (participants affected / at risk) | 24/43 | 45/84 | 46/85 | 44/85 | 30/43 | 28/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 24 mg s.c. q4w (N=43) | QGE031 72 mg s.c. q4w (N=84) | QGE031 240 mg s.c. q4w (N=85) | Omalizumab 300 mg s.c. q4w (N=85) | Placebo s.c. q4w (N=43) | QGE031 120 mg s.c. s.d. (N=42)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colon dysplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 24 mg s.c. q4w (N=43) | QGE031 72 mg s.c. q4w (N=84) | QGE031 240 mg s.c. q4w (N=85) | Omalizumab 300 mg s.c. q4w (N=85) | Placebo s.c. q4w (N=43) | QGE031 120 mg s.c. s.d. (N=42)
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 5 | 6 | 2 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 5 | 2 | 1
Injection site erythema (General disorders) | 0 | 2 | 5 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 3 | 6 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 5 | 1 | 0
Influenza (Infections and infestations) | 1 | 4 | 4 | 5 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 7 | 10 | 10 | 6 | 9
Urinary tract infection (Infections and infestations) | 0 | 5 | 4 | 5 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 7 | 13 | 17 | 17 | 13 | 10
Blood creatinine increased (Investigations) | 1 | 3 | 3 | 2 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1 | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 3
Dizziness (Nervous system disorders) | 2 | 5 | 2 | 2 | 4 | 0
Headache (Nervous system disorders) | 7 | 9 | 7 | 12 | 7 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 5 | 4 | 2 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 9 | 3 | 4 | 5 | 7
Hypertension (Vascular disorders) | 1 | 5 | 2 | 2 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.